CLINICAL TRIAL: NCT00038818
Title: CD8 Depleted Donor Lymphocyte Infusions for Patients With Relapse Or Residual Disease Following Allogeneic Stem Cell Transplantation
Brief Title: CD8 DLI for Patients With Relapse or Residual Disease Following Allogeneic Stem Cell Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Eligix (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-335
Record Dates: First submitted 2002-06-05; First posted 2002-06-07 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Myelogenous Leukemia; Multiple Myeloma; Non Hodgkin's Lymphoma; Hodgkin's Disease; Chronic Lymphocytic Leukemia
Keywords: CML; MM; NHL; HD; CLL; CD8 Depleted; Donor Lymphocyte
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CD8 DLI (Experimental): CD8 depleted DLI (Depleted Donor Lymphocyte Infusions)
  Interventions: Biological: CD8 Depleted Donor Lymphocyte

INTERVENTIONS:
Biological: CD8 Depleted Donor Lymphocyte

SUMMARY:
Primary Objectives:

To evaluate response rates of acute or chronic Graft-versus-host disease (GVHD) following CD8 depleted DLI (Depleted Donor Lymphocyte Infusions) in patients with Chronic myelomonocytic leukemia (CMML), chronic lymphoid leukemia (CLL), Non-Hodgkin's lymphoma (NLM), Multiple Myeloma (MM) and Hodgkin's Lymphoma (HD).

Secondary Objectives:

* To evaluate safety and treatment related mortality after CD8 depleted DLI.
* To evaluate the time to onset of GVHD following DLI and response to GVHD treatment.
* To evaluate the incidence and timing of pancytopenia following DLI.
* To evaluate disease-free survival, overall survival and relapse rates in three cohorts of patients; early relapse CML, late relapse CML and lymphoproliferative disorders (HD, CLL, NHL and MM).
* To evaluate the need and efficacy of second or subsequent CD8 depleted donor lymphocyte infusions.
* To evaluate the number of apheresis procedures needed to collect appropriate doses of CD4+ cells.

ELIGIBILITY:
* Patients of any age who have previously undergone allogeneic hematopoietic transplantation and have evidence of donor cell engraftment (>20% donor cell within three months of study entry)
* Expected survival >4 weeks
* CML patients with molecular, cytogenetic or hematologic relapse following allogeneic transplantation

  1. Molecular relapse- patients are eligible if bcr/abl is detectable at any time after day 180 post-allogeneic transplantation or if a negative bcr/abl PCR test was documented post-transplantation and the bcr/abl test is now positive by consecutive PCR determinations at least 4 weeks apart.
  2. Cytogenetic relapse-patients are eligible if standard cytogenetics demonstrate >10% t (9,22) positive cells greater than 60 days after myeloablative transplantation or 10% t (9,22) positive cells greater than 100 days after nonmyeloablative transplantation.
* CML patients with accelerated phase or blast crisis following allogeneic transplantation
* Patients with CLL, NHL, MM, or HD who have evidence of disease relapse or persistent disease at 60 days post-allo BMT and/or:

  1. MM- patients with a rising M-protein is detectable at 180 days post-transplant
  2. NHL - patients with molecular evidence of disease (bcl-2, t (4,11), etc.) at 180 days post transplant
  3. CLL, NHL or HD - patients with clear cut evidence of tumor growth at any time post-transplant are eligible
* Patients undergoing an HLA -identical or 5/6 antigen match transplant from a related or unrelated donor
* Patient's original donor must be available for lymphocyte donation
* There must be no evidence of active acute or graft-versus-host disease and patients should be off all immunosuppressive agents for, at least, two weeks prior to DLI. Patients on stable dose of methylprednisolone (<16 mg/d) without evidence of active GVHD are also eligible.
* Patients must have a Zubrod PS<2 (see appendix 7), Cr<2.5, bilirubin <3, and transaminases (SGPT, SGOT) <4x normal
* Patient must be able to sign informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2001-05; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Patient Response Rates of Acute or Chronic GVHD | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard Champlin, MD, BS, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org